CLINICAL TRIAL: NCT01395550
Title: Secondary Prevention Treatment in Patients Who Have Suffered a Cardiovascular Event.
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-CZA-XXX-2011/1
Record Dates: First submitted 2011-06-14; First posted 2011-07-15 (Estimated); Last update posted 2011-08-30 (Estimated); Status verified 2011-08

CONDITIONS: Cardiovascular Events

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
AstraZeneca was interested in knowing how Cardiologists and Physicians treat patients who have suffered a cardiovascular event.

ELIGIBILITY:
Inclusion Criteria:

* All patients who has experienced cardiovascular events

Exclusion Criteria:

* Patients with no cardiovascular events.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with cardiovascular events
Sampling Method: Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2010-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)